CLINICAL TRIAL: NCT00890539
Title: Methacholine Challenge: Comparison of Doubling and Quadrupling Methacholine Dose Regimes Using the Tidal Volume Method
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Saskatchewan (Other)
Responsible Party: Dr. Donald Cockcroft, University of Saskatchewan
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Diagnostic
Other Study IDs: BMC08-247
Record Dates: First submitted 2009-03-02; First posted 2009-04-30 (Estimated); Last update posted 2009-11-25 (Estimated); Status verified 2009-11

CONDITIONS: Asthma
MeSH Terms: conditions — Asthma

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Quadrupling (Experimental): methacholine challenge using quadrupling concentrations
  Interventions: Drug: Methacholine challenge
- doubling (Active Comparator): doubling concentrations of methacholine
  Interventions: Drug: Methacholine challenge

INTERVENTIONS:
Drug: Methacholine challenge — Clinical and research test used in asthma

SUMMARY:
The purpose of this study is to determine the difference (if any) in the result of the methacholine challenge (a test used by physicians in diagnosing asthma) when concentrations of methacholine are quadrupled versus doubled.

DETAILED DESCRIPTION:
The purpose of this study is to confirm that the tidal volume technique of methacholine delivery may be employed in methacholine challenges using a quadrupling dose schedule instead of the standard doubling dose schedule with similar diagnostic efficacy, with no increase in patient adverse events, and with a shorter investigational duration. This has previously been shown to be true using the dosimeter technique of methacholine challenge.

ELIGIBILITY:
Inclusion Criteria:

* You must be over 18 years of age; and
* You must have a diagnosis of asthma; and
* Excluding asthma, you are not aware of any other lung conditions or diseases.

Exclusion Criteria:

* You have a known hypersensitivity (i.e. an overreaction of your immune system) to methacholine or other parasympathomimetic agents or cholinesterase inhibitors (i.e. agents that act in a similar way via your nervous system - to be discussed with study personnel); or
* You are a nursing mother or if you are a woman of child bearing potential who is, may be, or intends to become pregnant during testing as the effects of methacholine inhalation in these situations are not known; or
* Your baseline lung function is poor (ie. your FEV or forced expiratory volume in one second, is less than 65% of your predicted values). This will be performed and explained by study personnel prior to commencing methacholine inhalation testing; or
* You have had any respiratory infections for the last four weeks; or
* If you have allergies, and have been exposed to agents that trigger your asthma within the last four weeks; or
* If you have any significant chronic medical condition.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Estimated)
Dates: Start 2009-02; Primary Completion 2009-03 (Actual); Study Completion 2009-03 (Actual)

PRIMARY OUTCOMES:
Methacholine PC20 | 1 week

SECONDARY OUTCOMES:
Subject measure of breathlessness - modified Borg scale | 1 week

CONTACTS AND LOCATIONS:
Overall Officials: Donald W Cockcroft, MD, Principal Investigator — University of Saskatchewan
Locations (1):
- University of Saskatchewan, Saskatoon, Saskatchewan, Canada